CLINICAL TRIAL: NCT04815707
Title: Surgical Repair Versus Expectant Management of Occult Inguinal Hernias: Strengthening the Evidence Base and Developing a Decision Tool
Brief Title: Treatment of Occult Inguinal Hernias
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Julie Holihan, Assistant Professor of Surgery-Clinical, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSC-MS-20-1327; KL2TR003168 (NIH)
Record Dates: First submitted 2021-03-02; First posted 2021-03-25 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Inguinal Hernia
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surgery (Other): Occult hernia found will be repaired at the same time as the initial inguinal hernia
  Interventions: Procedure: Occcult hernia repair
- Expectant Management (No Intervention): No surgery will be done if an occult hernia is found during the initial inguinal hernia surgery

INTERVENTIONS:
Procedure: Occcult hernia repair — The occult hernia will be repaired during the same inguinal hernia repair
  Arms: Surgery

SUMMARY:
Inguinal hernias are a common surgical problem. Best management of occult inguinal hernias, defined as hernias unable to be felt on physical exam, is unknown. From prior studies we know that most inguinal hernias will eventually become symptomatic and require surgery (70%). However, doing a repair on a very small, occult hernia may open the patient up to surgical complications, like chronic pain, earlier than necessary. This will be a multi-center randomized controlled trial of surgical repair versus expectant management of occult inguinal hernias. Patients undergoing laparoscopic unilateral inguinal hernia repair will be included. At the time of surgery, the surgeon will determine if there is an occult hernia contralateral side. If present, patients will be randomized to repair of the occult side or expectant management of the occult side. After 1 year post-operative data has been assessed, a decision tool will be created and administered to patients to aid in their decision making about treatments for their hernia.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Patients undergoing unilateral laparoscopic inguinal hernia repair, found to have a contralateral occult inguinal hernia

Exclusion Criteria:

* Patient has life expectancy of less than 2 years
* Patients unlikely to follow-up (e.g. live out of state, unable to be reached by phone/e-mail
* Non-English and Non-Spanish speakers
* Pregnant or breast-feeding patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Actual)
Dates: Start 2021-10-22 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Patient threshold value for need for future surgery in order to accept Expectant Management (EM) of an Occult Inguinal Hernia (OIH) determined using standard gamble technique | From Baseline up to 2 years post-operative
  Assessed by using a decision tool (standard gamble method) that will be developed using information gathered at 1 year post-operative

SECONDARY OUTCOMES:
Number of patients who develop any surgical complication | 30 days post-operative
  Includes: Wound complications (e.g. SSI, seroma, hematoma, wound dehiscence), complications with the mesh, and hospital readmissions
Hernia recurrence | 2 years post-operative
  recurrence of hernia
Operative re-intervention | 1 years post-operative
  Number of patients who had to have another surgery to repair their hernia
Assessment of chronic pain | 1 year post-operative
  Pain assessed by a validated visual assessment score
Progression of hernia signs or symptoms | 1 year post-operative
  Will be assessed by the physician during the 1 year post-operative abdominal exam visit
Change in Abdominal wall quality of life (AW-QOL) | From Baseline up to 2 years post-operative
  Hernia-related Quality of Life Survey (HerQLes) will be used to assess this. Consists of 12 statements that the patient will rate how much he/she agrees with each statement. They will rate each statement from 1 (Strongly Disagree) to 10 (strongly agree). These 12 ratings will be combined to form one score.
Number of patients with an occult inguinal hernia | Time of surgery
  Prevalence of patients found to have an occult inguinal hernia during their initial inguinal surgery
Groin pain on occult hernia side | 1 month and 1 year post-operative
  Pain assessed by a validated visual assessment score
Time duration for surgery | Time of surgery
  Assessed by looking at the total time for the surgery to repair the inguinal hernia(s)
Time off work due to the hernia surgery | Baseline to 2 years post-operative
  The amount of time (days) patients had to take time off from work for the hernia surgery
Time to resume normal activity from any hernia surgery | Baseline to 2 years post-operative
  The amount of time (days) it took for patients to resume their normal activities following hernia surgery
Satisfaction with Decision Scale | Baseline to 2 years post-operative
  A decision scale looking at risk vs. benefit of hernia surgery will be done with patients

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Lyndon B. Johnson General Hospital, Houston, Texas
  - Memorial Hermann Hospital-MIST Clinics, Houston, Texas